CLINICAL TRIAL: NCT03491059
Title: Feasibility of PET/CT to Detect the Oral/Pulmonary Distribution of Nicotine Following E-cigarette Use
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Michael V Knopp MD PhD, Professor, University of Cincinnati
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SP0232/2017H0463
Record Dates: First submitted 2018-02-21; First posted 2018-04-09 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: E-cigarette Use
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Full Study - Radiation (Experimental)
  Interventions: Drug: C-11 labeled nicotine; Radiation: PET/CT imaging
- Dress Rehearsal Only - No Radiation (No Intervention)

INTERVENTIONS:
Drug: C-11 labeled nicotine — Participants will vape with e-cigarettes radio-labeled with C-11 nicotine.
  Arms: Full Study - Radiation
Radiation: PET/CT imaging — After vaping with radio-labeled e-cigarettes, participants will be PET/CT imaged.
  Arms: Full Study - Radiation

SUMMARY:
The investigators aim to (1) establish a methodology for the evaluation of the biodistribution of radio-labeled nicotine following e-cigarette use, (2) determine the oral/pulmonary distribution of nicotine following e-cigarette use, and (3) determine the lowest required dose using the new digital PET/CT technology to provide detailed or accurate oral/pulmonary distribution data following e-cigarette use. Potential participants will be identified using advertisements such as brochures and online social media postings. After participants are identified, their eligibility will be determined using survey tools. All eligible participants will first have a screening visit at the WCIBMI for study participation. During this initial visit, subjects will be informed about the study in detail, and the relevant consent form will be reviewed and signed. If the participant agrees to participate, they will go through a full dress rehearsal. Up to 10 volunteers will only participate in the dress rehearsal. All other volunteers (30) will have a dress rehearsal without radiation exposure on day 1, and then on a second day, they will participate in the full imaging study using 11C-nicotine. During the imaging study, S-nicotine will be labeled with 11C and placed in the cartridge of an e-cigarette. There will be two dose groups: (A) 3 mCi dosage or (B) 9 mCi doses. The investigators intend to use dose level A; however, if it does not lead to the expected results, an alternate dose level as an option is needed, which is the 9 mCi (B) dose level. Subjects will take a maximum of 10 puffs (1 puff per 30 seconds) from the e-cigarette while positioned in the PET/CT system. Dynamic PET/CT imaging will be performed for a maximum of 60 minutes following inhalation. The subject will be placed in the PET camera in order to generate axial images of the following regions: head/neck (e.g., brain, oral cavity, and throat) and thorax (e.g., trachea, lungs). From the PET/CT images, quantitative radioactivity deposition will be determined, and the biodistribution and uptake/clearance will be evaluated. PET data will be acquired in listmode and subsequently used for simulation to determine the potentially lowest dose feasible using the next generation digital PET/CT technology.

DETAILED DESCRIPTION:
E-cigarette manufactures claim that e-cigarettes are safer than conventional cigarettes and that they may aid in smoking cessation. As a result, e-cigarettes are gaining popularity and use in the general public as a replacement for traditional cigarettes. However, little is known about the benefits and health risks of e-cigarette use. Although e-cigarettes have been shown to have negligible effect on carbon monoxide exposure and heart rate, they contain a variety of glycerols mixed with variable concentrations of nicotine. In addition, other substances are present in the refill solutions and/or resulting vapor, such as tobacco specific nitrosoamines, cotinine, aldehydes, metals, volatile organic compounds, tobacco alkaloids, and other pharmacologically active ingredients (although in concentrations much lower than in combustible traditional cigarettes). In addition, studies have shown that during the atomization process, there is a large range in the size of the particulate matter formed that is dependent upon both the device and refill solution used. It is well know that inhaled particulate matter may induce inflammation and may eventually lead to an increase in a variety of health risks including cardiovascular disease and emphysema. Although e-cigarettes are not currently regulated, studies have indicated that the e-liquid products should be regulated to ensure consistent nicotine delivery and to prohibit the use of ethylene glycol and other excipients that currently may be present at potentially harmful levels (high risk category). Additionally, only minimal valid data is available related to the biodistribution (deposition of nicotine and/or aerosol excipients) following inhalation. The evaluation of nicotine and aerosol deposition in the body will help to determine if the particulates formed during the atomization process may induce any serious health risks. Additionally, this data may be compared to traditional cigarette smoking to determine if e-cigarettes are truly a safer alternative to conventional cigarettes. In order to provide this data, quantitative methods need to be developed that allow for accurate in vivo biodistribution determination following inhalation.

To determine eligibility, participants will sequentially complete two eligibility surveys that include questions related to their use of e-cigarettes, tobacco cigarettes, other tobacco products, and pharmaceuticals. The brochures and social media postings will include a link to Eligibility Survey 1. Survey 1 will collect sensitive, medical information, but will be completely anonymous. Medical information will be collected solely for the purposes of determining participant eligibility and will be unlinked from any identifying participant information as well as future collected study data. Once participants are determined eligible by Survey 1, they will be directed to complete Survey 2 to confirm their eligibility. Survey 2 will ask participants questions about their vaping habits. If they are confirmed eligible from the survey, they will also be asked to provide their name and contact information (e-mail). Study personnel will then contact eligible participants to schedule a time for them to come to the WCIBMI for their initial visit. Responses from Survey 1 and Survey 2 will be completely unlinked to maintain anonymity about participants' medical information. Once the participant has been deemed eligible and indicated interest in participation, they will be invited to the WCIBMI to see the facilities, and the relevant consent form will be reviewed and signed. Participants will either participate solely in a dress rehearsal of the study, or they will participate in both a dress rehearsal and the full imaging study. During the dress rehearsal, participants will walk through the study process without the use of the 11C-nicotine e-cigarette and without performing any imaging. The participant will first disrobe and change to hospital scrubs. The subject will also wear full-body disposable personal protective equipment (PPE) including a gown, hairnet, double latex gloves, and foot coverings. Then, the subject will lay on the bed of the PET/CT imaging system and practice puffing in the supine position, the proper posture for PET scanning, and exhaling into the gas traps. Participants who are only participating in the dress rehearsal will use their own, personal e-cigarette to vape in the system. For participants who are participating in the full study, the investigators will provide them with the e-cigarette that they will use in the full study. Urine will be collected from female participants of the full study to confirm that they are not pregnant. During the study, first, S-nicotine will be labeled with C11 and placed in the cartridge of an e-cigarette. The S-nicotine may be given in two different doses. The investigators will focus on the 3 mCi C11 (Dose Level A) in the e-cigarette at the time of initial inhalation previously purified by HPLC. If 3 mCi does not yield adequate image quality, the dosage will be increased to 9 mCi (Dose Level B) for subsequent participants. To determine the appropriate dose level, the imaging scans will be reviewed independently at a minimum by three experienced investigators (Michael V. Knopp, Chadwick Wright, and Jun Zhang). Once the C11 labeled e-cigarette enters the facility, it may be placed in the dose calibrator for secondary dose confirmation and then transported directly to the imaging room. The subject will then be instructed to start inhalation (maximum 10 puffs at 30 second intervals) while positioned in the PET/CT system. Afterwards, the e-cigarette will be removed from the imaging system by a staff member, and the remaining activity of the E-liquid will be determined using a dose calibrator. PET/CT imaging will then be performed for a maximum of 60 minutes following inhalation. The subject will be placed in the PET camera as to generate axial slices in the following sectors: the brain, oral cavity, throat, and lungs. From the PET/CT images, quantitative radioactivity deposition will be determined, and the biodistribution and uptake/clearance will be evaluated. Acquired data will be used for listmode based simulation to determine the potentially lowest dose feasible using new digital PET/CT technology. After scanning, the subject will be removed from the imaging suite and will be asked to stay in the patient waiting/recovery area for up to 120 minutes (2 hours). Prior to release, the subject will be surveyed to ensure that any exhaled/emitted air is at background levels with respect to radiation. Additionally, all subjects will be contacted within 12 to 48 hours after release from the study to ensure that they are feeling well and have not experienced any adverse reaction to the study. Any adverse reactions will be recorded and reported immediately to the PI.

ELIGIBILITY:
Inclusion Criteria:

* males and females greater than or equal to 18 years of age
* current regular user of e-cigarettes (use at least once daily for the past 30 days) with nicotine strength > 6mg/ml
* health medical history
* abstinent from any tobacco/nicotine use for 4 hours prior to imaging

Exclusion Criteria:

* not a regular user of e-cigarettes
* pregnant or lactating (only excluded from imaging study)
* prisoner
* incapable of giving informed consent
* unable to lie flat on the scanner for extended periods of time
* unstable medical condition like heart disease, uncontrolled hypertension, thyroid disease, diabetes, renal or liver impairment, or glaucoma
* prostatic hypertrophy, stroke, or ulcer in past year
* psychiatric conditions such as schizophrenia, adult ADHD, or bipolar disorder
* current or regular use of psychiatric medications such as tranquilizers, antipsychotics, and/or antidepressants
* use of medications that are inducers of CYP2A6 (a nicotine metabolizing enzyme) such as rifampicin, dexamethasone, phenobarbital, and other anti-convulsant drugs
* unable to communicate in English
* current use of smokeless tobacco, tobacco cigarettes (5 and fewer a day)
* occasional use of pipes is permitted if subject abstains for the week prior to the study
* older than 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-16 (Estimated)

PRIMARY OUTCOMES:
Nicotine biodistribution | Up to 5 - 10 minutes
  We will measure the intensity of C11 labeled nicotine uptake, measured as SUV in different target and organ systems
Nicotine uptake | Up to 5 - 10 minutes
  We will measure the intensity of C11 labeled nicotine uptake, measured as SUV in the oral cavity, lungs, blood stream and brain
Nicotine clearance | Up to 5 - 60 minutes
  We will use the intensity of C11 labeled nicotine uptake, measured as SUV in the different target and organ systems in the PET imaging field of view and assess the change of uptake over time as a measure of its elimination

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Knopp, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

DOCUMENTS (1):
  • Study Protocol (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT03491059/Prot_000.pdf